CLINICAL TRIAL: NCT03781453
Title: POWERPLAY: Building Employee Health and Safety Through Prevention in Male-dominated Workplaces
Brief Title: POWERPLAY Phase 2: Development and Evaluation in Male-dominated Workplaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joan Bottorff (Other)
Collaborators: University of British Columbia (Other); Athabasca University (Other); University of Alberta (Other); Newcastle University (Other); University of Melboune (Unknown); University Technology Sydney (Unknown)
Responsible Party: Sponsor-Investigator, Joan Bottorff, Professor and Director of the Institute for Healthy Living and Chronic Disease Prevention, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 095244772
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Men; Health Behavior; Mental Health Wellness 1; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Health Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, pre-post study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: POWERPLAY — Employees from participating worksites will be invited to completed surveys prior to and following implementation of a workplace wellness program (called "POWERPLAY")

SUMMARY:
With funding from the Alberta Ministry of Labour (Grant #095244772), a program called POWERPLAY (www.powerplayatwork.com), designed to promote men's health at work, will be evaluated in workplaces in Alberta.

DETAILED DESCRIPTION:
In year 1, this project includes two main research components: 1. A pragmatic (real world) study will be conducted employing a quasi-experimental (not a randomized controlled trial), before and after design to evaluate the effectiveness of the POWERPLAY program. 2. An integrated set of research activities (systematic review, sleep behaviors and consultation groups) will be used to provide the basis for developing recommendations for promoting sleep health in male-dominated workplaces, and inform the development and testing of a POWERPLAY sleep health module (REST-UP) in Year 2.

ELIGIBILITY:
Inclusion Criteria:

* Men employed in participating workplaces, full-time or part-time, in any position within the organizations.

Exclusion Criteria:

* Although females may participate in the POWERPLAY program and surveys, they will not be included in the evaluation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility based on self-representation of gender identity
Enrollment: 498 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Moderate to Vigorous Physical Activity | 4 months
  Minutes of Moderate to Vigorous physical activity will be assessed using self-report at baseline and follow-up using the Godin Leisure-Time Exercise Questionnaire (Godin & Shephard, 1985). The Godin Leisure-Time Exercise Questionnaire contains three self-report questions that assess both the average frequency and duration (in minutes) of mild, moderate, and vigorous activities during free time over a typical week. Frequency and minutes are multiplied to obtain minutes per week (range from 0 and up). Weekly moderate and vigorous activity minutes will be summed and compared from baseline to follow-up, with higher scores indicating more activity. In addition, a cutoff of 150 minutes in 7 days will be used to classify participants as meeting or not meeting Canadian guidelines for physical activity at baseline and follow-up.
Mental Wellness | 4 months
  Mental well-being will be assessed using the well validated Short Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS) (Haver, Akerjordet, Caputi, Furunes, & Magee, 2015; Tennant et al., 2007) at baseline and follow-up. Participants respond to 7-items (e.g., "I've been feeling optimistic about the future") on a 5-point Likert scale ranging from none of the time (1) to all of the time (5), with higher scores reflecting greater mental well-being. The SWEMWBS is scored by summing the score for each of the seven items (possible range 7-35).

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Shell Canada Ltd (Scotford Site), Ft Saskatchewan, Alberta
  - Roper Ventures, Rocky Mountain House, Alberta
  - PeroxyChem, Prince George, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: POWERPLAY program website — http://www.powerplayatwork.com/